CLINICAL TRIAL: NCT03850379
Title: Ciprofloxacin Versus Levofloxacin and Rate of Breakthrough Infections in Hematopoietic Stem Cell Transplant Patients
Brief Title: Ciprofloxacin Versus Levofloxacin in Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12124)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Prophylaxis; Stem Cell Transplant Complications
MeSH Terms: interventions — Levofloxacin; Ciprofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levo (Experimental): Levofloxacin 500 mg once daily
  Interventions: Drug: Levofloxacin
- Cipro (Active Comparator): Ciprofloxacin 500 mg BID
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Levofloxacin — This is a prospective study comparing consecutive patients who will be be receiving ciprofloxacin prophylaxis vs. levofloxacin prophylaxis for Stem cell transplant till engraftment defined as ANC >1000
  Arms: Levo
Drug: Ciprofloxacin — This is a prospective study comparing consecutive patients who will be be receiving ciprofloxacin prophylaxis vs. levofloxacin prophylaxis for Stem cell transplant till engraftment defined as ANC >1000
  Arms: Cipro

SUMMARY:
Ciprofloxacin and levofloxacin are both in guidelines to use for prophylaxis in autologous and allogeneic Stem cell transplant.Ciprofloxacin was recently replaced by levofloxacin as the preferred agent in some transplant centers. In some small retrospective studies ciprofloxacin prophylaxis was associated with a higher rate of breakthrough gram positive bloodstream infections. However, the optimum oral agent for antibacterial prophylaxis in transplant recipients remains uncertain.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-75 years of age with a diagnosis of a hematological malignancy. Meet the stem cell transplant program criteria to undergo autologous or allogeneic hematopoietic stem cell transplantation.

Exclusion Criteria:

* Prolonged QT
* Allergies to ciprofloxacin or levofloxacin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford, Detroit, Michigan, United States

REFERENCES:
- [Result] Farhan S, Mazur I, Hartzell S, Xie P, Neme K, German A, Mikulandric N, Patel K, Wu M, Kortam N, Yaseen A, Sweidan A, Latack K, Emole J, Peres E, Abidi MH, Ramesh M. Ciprofloxacin versus levofloxacin prophylaxis in hematopoietic stem cell transplantation: A randomized trial. Int J Infect Dis. 2024 Oct;147:107172. doi: 10.1016/j.ijid.2024.107172. Epub 2024 Jul 15. PMID 39019103

RESULTS

PARTICIPANT FLOW:
Groups:
- Levo: Levofloxacin 500 mg once daily
  Levofloxacin: This is a prospective study comparing consecutive patients who will be be receiving ciprofloxacin prophylaxis vs. levofloxacin prophylaxis for Stem cell transplant till engraftment
- Cipro: Ciprofloxacin 500 mg BID
  Ciprofloxacin: This is a prospective study comparing consecutive patients who will be be receiving ciprofloxacin prophylaxis vs. levofloxacin prophylaxis for Stem cell transplant till engraftment
Period: Overall Study
Arm/Group | Levo | Cipro
Started | 154 | 154
Completed | 154 | 154
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levo | Cipro | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [55 to 68] | 62 [54 to 69] | 63 [54 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 66 | 136
  Male | 84 | 88 | 172
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 93 | 100 | 193
  African Americans | 50 | 41 | 91
  Others | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 154 | 154 | 308

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Bloodstream Bacterial Infections
Description: to assess proportion of bloodstream bacterial infections in the ciprofloxacin group compared to levofloxacin group up to day 60 after stem cell transplant
Time Frame: 60 days post stem cell transplant
Measure: Number; unit: participants
Arm/Group | Levo | Cipro
Number analyzed (Participants) | 154 | 154
participants | 18 | 18

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Levo | Cipro
All-Cause Mortality (participants affected / at risk) | 42/154 | 54/154
Serious Adverse Events (participants affected / at risk) | 23/154 | 20/154
Other Adverse Events (participants affected / at risk) | 0/154 | 0/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levo (N=154) | Cipro (N=154)
arrythmias (Cardiac disorders) | 16 | 12
fluid overload (Cardiac disorders) | 3 | 1
encephalopathy (Nervous system disorders) | 2 | 1
seizure (Nervous system disorders) | 0 | 1
bowel obstruction (Gastrointestinal disorders) | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
syncope (Cardiac disorders) | 0 | 1
CMV viremia (Infections and infestations) | 0 | 1
hematoma (Blood and lymphatic system disorders) | 0 | 1
thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Our study has several limitations that need to be considered when interpreting the results. First, the study was randomized but open-label. This could have influenced decisions about patient care, potentially biasing the results. Second, the study only documented infections until day 60, which might not capture resistant bacterial infections that may occur later. Third, this study unfortunately lacks information on the gut microbiome, which might play a role in the observed outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03850379/Prot_SAP_001.pdf